CLINICAL TRIAL: NCT03199339
Title: Phase 1, Partially-Blind, Placebo Controlled Randomized, Combined SAD With Food Effect Cohort and MAD and DDI Study to Evaluate Safety, Tolerability, PK and PK Interaction Between TBA-7371 With Midazolam and Bupropion in Healthy Subjects.
Brief Title: A Phase 1 Study to Evaluate Safety, Tolerability, PK, and PK Interactions of TBA-7371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TBA-7371-CL001
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-02

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: tuberculosis; TBA7371; TBA-7371; TB Alliance; TB; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Midazolam; Bupropion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Part 1 and Part 2 participants will be masked, Part 3 participants will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- SAD Part 1 Cohort 1 First Dose - Active (Active Comparator): N = 2, 100 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 1 First Dose - Placebo (Placebo Comparator): N = 1, 100 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- SAD Part 1 Cohort 1 Second Dose - Active (Active Comparator): N = 4, 100 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 1 Second Dose -Placebo (Placebo Comparator): N = 1, 100 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- SAD Part 1 Cohort 2 - Active (Active Comparator): N= 6, 250 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 2 - Placebo (Placebo Comparator): N = 2, 250 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- SAD Part 1 Cohort 3 - Active (Active Comparator): N = 6, 500 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 3 - Placebo (Placebo Comparator): N = 2, 500 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- SAD Part 1 Cohort 4 - Active (Active Comparator): N = 6, 1000 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 4 - Placebo (Placebo Comparator): N = 2, 1000 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- SAD Part 1 Cohort 5 - Active (Active Comparator): N = 6, 1500 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- SAD Part 1 Cohort 5 - Placebo (Placebo Comparator): N = 2, 1500 mg TBA-7371 or matching placebo
  Interventions: Drug: Placebo
- MAD Part 2 Cohort 1 - Active (Active Comparator): N = 9, 100 mg TBA-7371 or matching placebo
  Interventions: Drug: TBA-7371
- MAD Part 2 Cohort 1 - Placebo (Placebo Comparator): N = 3, 100 mg TBA-7371 or matching placebo for 14 days
  Interventions: Drug: Placebo
- MAD Part 2 Cohort 2 - Active (Active Comparator): N = 9, 200 mg TBA-7371 or matching placebo for 14 days
  Interventions: Drug: TBA-7371
- MAD Part 2 Cohort 2 - Placebo (Placebo Comparator): N = 3, 200 mg TBA-7371 or matching placebo for 14 days
  Interventions: Drug: Placebo
- MAD Part 2 Cohort 3 - Active (Active Comparator): N = 9, 400 mg TBA-7371 or matching placebo for 14 days
  Interventions: Drug: TBA-7371
- MAD Part 2 Cohort 3 - Placebo (Placebo Comparator): N = 3, 400 mg TBA-7371 or matching placebo for 14 days
  Interventions: Drug: Placebo
- DDI Part 3 Cohort 1 (Active Comparator): 14 subjects to receive midazolam and bupropion before and after orally giving 200mg of TBA-7371, 1 per day for 14 days
  Interventions: Drug: TBA-7371

INTERVENTIONS:
Drug: TBA-7371 — The test product is TBA-7371 25 mg/ml oral suspension formulation and TBA-7371 matching placebo oral suspension.
  Other Names: Midazolam (oral syrup); Bupropion
  Arms: DDI Part 3 Cohort 1; MAD Part 2 Cohort 1 - Active; MAD Part 2 Cohort 2 - Active; MAD Part 2 Cohort 3 - Active; SAD Part 1 Cohort 1 First Dose - Active; SAD Part 1 Cohort 1 Second Dose - Active; SAD Part 1 Cohort 2 - Active; SAD Part 1 Cohort 3 - Active; SAD Part 1 Cohort 4 - Active; SAD Part 1 Cohort 5 - Active
Drug: Placebo — The test product is TBA-7371 25 mg/ml oral suspension formulation and TBA-7371 matching placebo oral suspension.
  Other Names: Matching Placebo for TBA-7371
  Arms: MAD Part 2 Cohort 1 - Placebo; MAD Part 2 Cohort 2 - Placebo; MAD Part 2 Cohort 3 - Placebo; SAD Part 1 Cohort 1 First Dose - Placebo; SAD Part 1 Cohort 1 Second Dose -Placebo; SAD Part 1 Cohort 2 - Placebo; SAD Part 1 Cohort 3 - Placebo; SAD Part 1 Cohort 4 - Placebo; SAD Part 1 Cohort 5 - Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single and multiple doses of TBA-7371 in healthy subjects

DETAILED DESCRIPTION:
Three - part, partially-blinded, placebo controlled, combined single ascending dose with a food effect cohort and multiple ascending dose and a drug-drug interaction study to be conducted in one study center in the United States.

Part 1 has a single ascending dose (SAD) design with up to 5 planned dose levels. Based on the interim PK for the dose escalation decisions, a dose cohort will be selected to return for an additional dose after a high calorie, high fat meal.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and PK assessment of TBA-7371. Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability and PK from the previous cohort has been demonstrated to permit proceeding to the next cohort.

Interim PK analyses will be performed for the dose escalation decisions, to select the intermediate dose for the food effect cohort, and to reconsider the sampling time points as the study progresses. All samples will be sent for analysis and the bioanalytical lab will be unblinded and only run the analysis on active treatment subjects. Data from the analysis used for the escalation meetings will only include active treatment subjects, and will be blinded by subject.

Subjects will be housed in the WCT clinic from at least 24 hours prior (from Day -2), until 48 hours after dosing. Subjects will return for subsequent follow up safety and PK assessments on Day 4 and will be contacted via a phone call for follow-up questioning about adverse events 7 days later (Study Day 11). One cohort will return after a washout of at least 7 days or five half-lives (whichever is longer) of their fasting dose to receive the same intermediate dose (TBD mg) under fed conditions.

Part 2 has a multiple ascending dose design. The dose cohorts for Part 2 will be determined based on model predictions to determine the steady-state Cmax exposure, and safety from Part 1.

In this multiple ascending dose part, each subject will be administered TBA-7371 or matching placebo for 14 days with corresponding PK measurements. Three dose cohorts are planned. After each dose cohort, the Sponsor and Investigator will review the PK and safety data before proceeding to the next dose level.

Part 3 has an open-label, multi-dose, fixed sequence drug-drug interaction study design. The dose of TBA-7371 to be studied will dependent on the interim PK analyses and safety from Part 2.

In this DDI part, each subject (n=14) will be administered midazolam (2 mg suspension) and bupropion (150 mg, tablet) together on Day 1, followed by a 7-day washout, followed by administration of TBA-7371 on Days 8 through 21, followed by administration of midazolam, and bupropion on Day 22. PK will be assessed for midazolam on Days 1 and 22, bupropion on Days 1 - 5 and 22 - 26, and TBA-7371 on Days 8-21.

At the end of Part 1 and at the end of Part 2, pharmacokinetic and safety data along with reasons for doses for the next part (Part 2 and Part 3, respectively) will be sent to the Food and Drug Administration (FDA) for review and approval. The study will not proceed to Part 2 or Part 3 until the FDA provides approval.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria and none of the exclusion criteria to be eligible for participation in the study, unless otherwise specified.

1. Healthy adult male and females of non-childbearing potential, 19 to 50 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) and a body weight of no less than 50.0 kg.
3. Medically healthy with no clinically significant screening results (e.g., laboratory profiles, medical histories, vital signs, ECGs, physical examination) as deemed by the Investigator.
4. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 6 months prior to dosing.
5. Females of non-childbearing potential, having undergone one of the following sterilization procedures at least 6 months prior to dosing:

   i. Hysteroscopic sterilization ii. Bilateral tubal ligation or bilateral salpingectomy iii. Hysterectomy iv. Bilateral oophorectomy v. or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum follicle stimulating hormone (FSH) levels consistent with postmenopausal status at screening.
6. Non-vasectomized males (or males vasectomized less than 120 days prior to study start), must agree to the following during study participation and for 90 days following the last administration of study drug:

   1. use a condom with spermicide while engaging in sexual activity or be sexually abstinent
   2. not donate sperm during this time. In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to study start.
7. Willing to answer inclusion and exclusion criteria questionnaire at check-in.
8. Subject understands study procedures and provides written informed consent for the trial.
9. Be able to comply with the protocol and the assessments therein, including all restrictions.
10. Is willing and able to remain in the study unit for the entire duration of the assigned confinement period and return for outpatient visits.
11. If enrolled in Part 1 and assigned to the fasted/fed cohort, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria at screening or check-in, as appropriate.

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as determined by the Investigator to be clinically relevant.
2. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. Surgery within the past 90 days prior to dosing as determined by the Investigator to be clinically relevant, or any history of cholecystectomy.
4. History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.
5. Female subjects who are pregnant or lactating.
6. Positive results for the urine drug/alcohol screen at screening or check-in.
7. Positive urine cotinine at screening or check in.
8. Serum magnesium potassium, or calcium laboratory values outside of the normal range at screening.
9. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
10. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening, Day -2 (check-in), Day -1, or predose. Out-of-range vital signs may be repeated once for confirmation.
11. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening, Day -2 (check-in), Day -1, or predose. Out-of-range vital signs may be repeated once for confirmation.
12. Any electrocardiogram abnormality at Screening (as deemed by decision of the Investigator and the Sponsor's Medical Monitor).

    NOTE: The following can be considered not clinically significant without consulting the Sponsor's Medical Monitor:

    i. Mild first degree A-V block (P-R interval <0.23 sec) ii. Right or left axis deviation iii. Incomplete right bundle branch block iv. Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
13. QTcF interval >450 msec for males or >470 msec for females at screening, Day -2, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome.
14. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
15. History of one or any combination of, the following:

    i. Seizures or seizure disorders ii. Brain surgery. iii. History of head injury in the last five years iv. Any serious disorder of the CNS or related neurological system, particularly one that may lower the seizure threshold.

    v. History of seizures
16. Use of any prescription medication within 14 days prior to dosing.
17. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing, except acetaminophen. Up to 3 grams per day of acetaminophen is allowed at the discretion of the Investigator prior to dosing.
18. Use of any drugs or substances known to be significant inhibitors of Cytochrome P450 (CYP) enzymes and/or significant inhibitors or substrates of P-glycoprotein (P-gp) and/or Organic anion transporting polypeptides (OATP) within 14 days prior to the first dose of study drug.
19. Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 30 days prior to the first dose of study drug.
20. Use of any drugs or substance known to lower the seizure threshold.
21. Blood donation or significant blood loss within 56 days prior to dosing.
22. Plasma donation within 7 days prior to dosing.
23. Participation in another clinical trial within 28 days prior to dosing. Consumption of foods and beverages containing the following substances will be prohibited
24. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
25. Unwilling to remove any artificial nails (e.g. acrylic, gel) or fingernail polish and not use such products for the duration of the study.
26. Is colorblind (assessed using the Ishihara Color Vision Test)

    Additionally, the following exclusion applies only to subjects in Part 1, the SAD study:
27. Is lactose intolerant.

    Additionally, the following exclusion applies only to subjects in Part 1 and 2, the SAD and MAD studies:
28. History or presence of allergic or adverse response to Listerine breath strips or aspartame.

    Additionally, the following exclusions apply only to subjects in Part 3, the DDI study:
29. History or presence of allergic or adverse response to midazolam, bupropion, or related drugs.
30. History of presence of acute narrow-angle or untreated open-angle glaucoma
31. Current or prior diagnosis of bulimia or anorexia nervosa
32. Abrupt discontinuation of alcohol, benzodiazepines, barbiturates, or anti-epileptic drugs within 14 days prior to the first dose of study treatment
33. Discontinued the use of monoamine oxidase inhibitors (MAOs) within 14 days prior to the first dose of study treatment
34. History or presence of suicidal ideation or suicidal behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS, Baseline/Screening Version) at the Screening Visit.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of TBA-7371 in healthy subjects by number and severity of treatment emergent adverse events (TEAEs) | Days 0-28 (depending on dosing schedule)
  The primary endpoint of the study will be the number and severity of treatment emergent adverse events (TEAEs) following single doses of TBA-7371 and placebo

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of single and multiple doses of TBA-7371 AUC(0-t) | Days 0-28 (depending on dosing schedule)
  This will be measured through AUC(0-t). AUC = Area under the curve, t = determined time point
Pharmacokinetics (PK) of single and multiple doses of TBA-7371 using Cmax | Days 0-28 (depending on dosing schedule)
  This will be measured through Cmax. , Cmax = maximum observed concentration
Pharmacokinetics (PK) of single and multiple doses of TBA-7371 using Tmax | Days 0-28 (depending on dosing schedule)
  This will be measured through Tmax, Tmax = Time of the maximum drug concentration (obtained without interpolation)
Compare the rate and extent of absorption of a single oral dose of TBA-7371 using AUC, when administered after a high-calorie, high-fat meal versus when it's administered fasting in healthy adult subjects | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like AUC; AUC = Area under the curve
Compare the rate and extent of absorption of a single oral dose of TBA-7371 using Cmax, when administered after a high-calorie, high-fat meal versus when it's administered fasting in healthy adult subjects | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like Cmax; Cmax = maximum observed concentration
Compare the rate and extent of absorption of a single oral dose of TBA-7371 using Tmax, when administered after a high-calorie, high-fat meal versus when it's administered fasting in healthy adult subjects | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like Tmax; Tmax = Time of the maximum drug concentration (obtained without interpolation)
Effects of multiple-dose administration of TBA-7371 on the pharmacokinetics of midazolam and bupropion using AUC | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like AUC; AUC = Area under the curve
Effects of multiple-dose administration of TBA-7371 on the pharmacokinetics of midazolam and bupropion using Cmax | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like Cmax; Cmax = maximum observed concentration
Effects of multiple-dose administration of TBA-7371 on the pharmacokinetics of midazolam and bupropion using Tmax | Days 0-28 (depending on dosing schedule)
  This will be measured through PK parameters like Tmax; Tmax = Time of the maximum drug concentration (obtained without interpolation)
Safety and tolerability of the combination of TBA7371 with midazolam and bupropion by the number and severity of treatment emergent adverse events (TEAEs) | Days 0-28 (depending on dosing schedule)
  The primary endpoint of the study will be the number and severity of treatment emergent adverse events (TEAEs) following single doses of TBA-7371 and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Del Parigi, MD, Study Director — Global Alliance for TB Drug Development
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States